CLINICAL TRIAL: NCT04172038
Title: SMART Stepped Care Management for Low Back Pain in the Military Health System
Acronym: SMART LBP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: University of Utah (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH); Madigan Army Medical Center (U.S. Federal Agency); 59th Medical Wing (U.S. Federal Agency); Tripler Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dan Rhon, DSc, PT, Physical Performance Service Line, Office of the Surgeon General, Brooke Army Medical Center
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 908761; 4UH3AT009763-03 (NIH)
Record Dates: First submitted 2019-11-18; First posted 2019-11-21 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain; Chronic Pain; Military Personnel; Veterans
Keywords: stepped care; physical therapy; mindfulness; holistic health; military medicine
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Randomization Trial (SMART) comparing the effectiveness and cost-effectiveness of Stepped Care pain management options, examining sequencing, and heterogeneity of effects in pre-specified subgroups.
Who Masked: Outcomes Assessor
Masking Description: 8-week and 18-week follow-up assessments will be performed by a research assistant who will be blind to participants' treatment group assignment. Participants will be reminded by the research assistant not to discuss aspects of their treatment during assessments. If a research assistant becomes unblinded during the course of a participants study participation, he or she will not be allowed to conduct additional follow-up assessments. Instances of unblinding during an assessment will be recorded as an unexpected event.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase I: Physical Therapy (PT) (Experimental): Initial Randomization: The initial PT treatment session will occur within 7 days of enrollment in the study. Precise dosage (i.e, number of PT sessions) will be at the discretion of the physical therapist directing the participant's care, up to a maximum of 2-3 sessions per week over the 6-week Phase I treatment period.
  Interventions: Behavioral: Physical Therapy
- Phase I: Move to Health (M2H) (Experimental): Initial Randomization: M2H is a key component of Army Medicine's "System for Health", along with the Performance Triad. It is a person-centered, holistic, and experience-centric approach to promoting healthy behaviors (nutrition, physical activity, sleep, instrinsic factors, extrinsic factors). Precise dosage (i.e, number of M2H sessions) will be at the discretion of the health coaches. Sessions may be delivered in-person or utilize technology including text messaging, telephone, e-mail, video chat, app-based self-management etc.
  Interventions: Behavioral: Move 2 Health (M2H)
- Phase II: Combine PT & M2H (Experimental): Sequential Randomization: Participants randomized to receive a combination of PT and M2H as a Phase II intervention will continue their Phase I treatment (either M2H or PT). The participant will begin the treatment component that was not part of their Phase I intervention.
  Interventions: Behavioral: Physical Therapy; Behavioral: Move 2 Health (M2H)
- Phase II: MORE Mindfulness (Experimental): Sequential Randomization: Participants randomized to receive mindfulness as a Phase II intervention will discontinue their Phase I treatment. The Mindfulness-Oriented Recovery Enhancement (MORE) treatment was designed specifically to address symptoms and underlying mechanisms of chronic pain in the military context and is led over 8 individual sessions.
  Interventions: Behavioral: MORE Mindfulness

INTERVENTIONS:
Behavioral: Physical Therapy — Physical therapy will be delivered using a guideline-concordant approach based off the Department of Defense -Veterans Affairs Low Back Pain Guidelines, focusing on risk-stratified care deliver (using the STarT Back tool as an adjunct).
  Other Names: physiotherapy
  Arms: Phase I: Physical Therapy (PT); Phase II: Combine PT & M2H
Behavioral: Move 2 Health (M2H) — Participants will receive education for self-management (video and written materials) to introduce the key domains of holistic health in the Move to Health (M2H) model and their relationship to chronic LBP. Next, the participant will complete a Personal Health Inventory. The Inventory will be reviewed by the health coach and patient in order to identify specific domains for priority based on patient preference:
  1. Sleep
  2. Physical Activity
  3. Nutrition
  4. Intrinsic Well-Being (Personal Development, Spiritual Well-Being, Emotional Well-Being)
  5. Extrinsic Well-Being (Family/Social Relationships, Surroundings)
  Care may range from guided self-management with the researcher to a specialist referral (e.g., sleep specialist, dietician, behavioral health provider, etc.).
  Arms: Phase I: Move to Health (M2H); Phase II: Combine PT & M2H
Behavioral: MORE Mindfulness — Throughout the intervention, three core areas are emphasized. Activities include exercises and at-home work for participants to reinforce these core areas.
  1. Mindfulness
  2. Cognitive reappraisal
  3. Savoring of positive experiences
  Arms: Phase II: MORE Mindfulness

SUMMARY:
This study will be sequential, randomization trial where patients with chronic low back pain are initially randomized to receive 1 of 2 treatments (physical therapy OR Move 2 Health). This will be Phase I of the study intervention. Patients who do not respond to treatment after 6 weeks will undergo a subsequent sequential randomization. This will be Phase II of the study intervention. Patients in Phase II will be randomized to receive 1 of 2 treatments (addition of physical therapy or Move 2 Health, whichever one they did not receive OR the MORE Mindfulness intervention). Patients will be followed for 1 year after enrollment.

DETAILED DESCRIPTION:
Improving non-pharmacologic management of chronic pain is a priority for the Military Health System (MHS) within the Department of Defense (DoD) and the most common chronic pain condition in the MHS and civilian healthcare is low back pain (LBP). Key questions exist however about the relative effectiveness of various strategies at different Steps, how to sequence treatments and individualize care based on specific patient characteristics and the resource implications. This study will recruit active duty military members or members of Reserves or National Guard on active duty, family members of active duty personnel, or Tricare beneficiaries seeing a primary care provider for chronic LBP in an MHS facility, ages 18-65. All participants will first receive 6 weeks of Phase I care with either physical therapy (PT) or Move to Health (M2H) interventions. After Phase I the investigators will assess response to initial treatment strategy. Phase I responders will be receive up to 2 additional sessions of treatment to facilitate a transition to self-management. Phase I non-responders will be randomly assigned to a more intensive Phase II treatment of either mindfulness or a combined PT+M2H intervention for 8 weeks. Randomization at each phase will be stratified by site, gender, and active duty status (adding Phase I treatment assignment at Phase II). Follow-up assessments for all participants will occur at 18 weeks (conclusion of Phase II), 6 months and 12 months after enrollment. Outcomes include patient-reported measures and health care costs.

ELIGIBILITY:
Inclusion Criteria:

1. Active duty military member (Army, Navy, Air Force, Marines) or member of Reserves or National Guard on active duty, a family member of active duty personnel, or Tricare beneficiary receiving care in a participating Military Treatment Facility.
2. Age 18 - 65 years at the time of enrollment.
3. Receiving Step 1 chronic LBP care based on VA Stepped Care Pain Management model defined as:

   a. Seen by a health care provider for chief complaint of LBP with or without symptoms into the buttocks or legs within past the 30 days.
   * Chief complaint of LBP which may be self-reported or identified by primary International Classification of Disease (ICD), 10th edition codes of LBP (M54.5, M54.9, S33.012), lumbar degenerative change (M51.36, M51.37, M48.06, M47.817), lumbar disc herniation/radiculitis (M54.16, M54.17, M51.26, M51.27, M54.3).
4. Meets NIH Task Force145 definition of chronic LBP based on two questions:

   How long has LBP has been an ongoing problem for you? and How often has LBP been an ongoing problem for you over the past 6 months? A response of greater than 3 months to question 1, and "at least half the days in the past 6 months" to question 2 is required to satisfy the NIH definition of chronic LBP.
5. Anticipates ability to attend treatment sessions over a 16 week period following enrollment with no planned absence of 2 weeks or more for training, vacation or any purpose.

Exclusion Criteria:

1. Signs of serious or systemic pathology as a cause of LBP including spine fracture, neoplasm, inflammatory disease (e.g., ankylosing spondylitis), vertebral osteomyelitis, etc.
2. Knowingly pregnant
3. Has received interventions for LBP that involves providers other than primary care in the past 6 months. This includes physical therapy or behavioral pain management or counseling as well as specialist physician consultations, chiropractic, etc.
4. Has received any interventional pain procedures (e.g., spinal injections), inter-disciplinary pain management, integrated chronic pain and substance use treatment programs, etc. in the past 6 months
5. Has received any lumbar spine surgery in the past year.
6. Retiring from active duty within 12 months, pending a medical evaluation board, discharge from the military for medical reasons, or pending or undergoing any litigation for an injury.
7. At elevated acute risk for suicide (i.e., risk is below the level requiring either consultation or urgent action based on Veterans Affairs-Department of Defense Clinical Practice Guideline for Assessment and Management of Patients at Risk for Suicide)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
PROMIS-Pain Interference Computer Adapted Test (PI-CAT) | 1 year
  Computer-adapted assessment using a 44-item bank measuring the self-reported consequences of pain on relevant aspects of life including impact on social, emotional, cognitive, physical and recreational activities. All Patient-Reported Outcomes Measurement Information System (PROMIS®) scores are reported on a T-score metric with a score of 50 points aligning with the general population mean and a standard deviation of 10. Higher scores indicate greater pain interference.

SECONDARY OUTCOMES:
PROMIS Physical Function Computer Adapted Test (PF-CAT) | 1 year
  Computer-adapted assessment using a 121-item bank measuring current, self-reported capability related to physical activities. All PROMIS scores are reported on a T-score metric with a score of 50 points aligning with the general population mean and a standard deviation of 10. Higher scores indicate greater physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Fritz, PhD, Principal Investigator — University of Utah; Daniel I Rhon, PhD, Principal Investigator — Brooke Army Medical Center
Locations (4):
- United States (4):
  - Desmond Doss Health Clinic, Schofield Barracks, Hawaii
  - Brooke Army Medical Center, San Antonio, Texas
  - Wilford Hall Ambulatory Surgical Center, San Antonio, Texas
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
There are plans to share data within the NIH-DoD-VA Pain Management Collaboratory (PMC) for future initiatives related to the PMC
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Depends on the timeline established by the PMC
Access Criteria: With reasonable request to the PI, and for any DHA-owned data, after following the established process by the Defense Health Agency to procure a Data Sharing Agreement.
URL: https://painmanagementcollaboratory.org/

REFERENCES:
- [Background] Main CJ, George SZ. Psychologically informed practice for management of low back pain: future directions in practice and research. Phys Ther. 2011 May;91(5):820-4. doi: 10.2522/ptj.20110060. Epub 2011 Mar 30. PMID 21451091
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Chou R, Huffman LH; American Pain Society; American College of Physicians. Nonpharmacologic therapies for acute and chronic low back pain: a review of the evidence for an American Pain Society/American College of Physicians clinical practice guideline. Ann Intern Med. 2007 Oct 2;147(7):492-504. doi: 10.7326/0003-4819-147-7-200710020-00007. PMID 17909210
- [Derived] Rhon DI, Fritz JM, Greenlee TA, Dry KE, Mayhew RJ, Laugesen MC, Dragusin E, Teyhen DS. Move to health-a holistic approach to the management of chronic low back pain: an intervention and implementation protocol developed for a pragmatic clinical trial. J Transl Med. 2021 Aug 18;19(1):357. doi: 10.1186/s12967-021-03013-y. PMID 34407840
- See also: VA/DoD Clinical Practice Guidelines for Diagnosis and Treatment of Low Back Pain (LBP) (2017) — https://www.healthquality.va.gov/guidelines/Pain/lbp/
- See also: NIH-DoD-VA Pain Management Collaboratory — https://painmanagementcollaboratory.org/smart-stepped-care/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT04172038/Prot_SAP_001.pdf
  • Informed Consent Form (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT04172038/ICF_000.pdf